CLINICAL TRIAL: NCT06224634
Title: The Effect of Anti-IL17 on Airway Hyperresponsiveness and Resistance: a Longitudinal Cohort Study
Brief Title: The Effect of Anti-IL17 on Airway Hyperresponsiveness and Resistance
Status: Recruiting | Type: Observational
Sponsor: Copenhagen University Hospital, Hvidovre (Other)
Responsible Party: Principal Investigator, Jonas Baekdal, Medical doctor, Copenhagen University Hospital, Hvidovre
Other Study IDs: AHR after Anti-IL-17
Record Dates: First submitted 2024-01-16; First posted 2024-01-25 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2024-08

CONDITIONS: Asthma
Keywords: Asthma; Interleukin 17; ankylosing spondylitis; Psoriasis; Airway hyperresponsiveness
MeSH Terms: conditions — Asthma; Spondylitis, Ankylosing; Psoriasis; Respiratory Hypersensitivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum and plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This observational longitudinal cohort study aims to assess the effect of monoclonal antibodies targeting interleukin 17 (anti-IL-17) on airway hyperreactivity and airway resistance. The study involves adult participants suffering from dermatological or rheumatological illness, who are planning to start treatment with monoclonal antibodies targeting interleukin 17 as a part of the treatment of these diseases.

The primary outcome of this study will be changes in airway hyperresponsiveness to methacholine challenge reported as response-dose-ratio before and after initiation of anti-IL17 treatment regardless of presence of respiratory disease. Furthermore, the potential effect of anti-IL-17 on airway resistance will be assessed using conventional spirometry for measuring changes in FEV1 and Airwave oscillometry.

A reduced degree of airway hyperreactivity and airway resistance after initiating ani-IL-17 could indicate effectiveness of anti-IL-17 in asthma patients which would have to be examined further in a population of asthma patients.

DETAILED DESCRIPTION:
Background:

Antibodies towards interleukin 17 (IL-17) are approved for treating various rheumatological and dermatological diseases like psoriatic arthritis, ankylosing spondylitis and plaque psoriasis. In recent years, IL-17 has been suggested as a potential driver of severe non-Type 2 asthma because of its' association with glucocorticoid resistance and symptoms of severe asthma. Since conventional treatment is often less effective in patients suffering from non-Type 2 asthma, sometimes adequate disease control cannot be achieved, thus limiting these patients' opportunity for physical exercise, and thereby increasing the risk of obesity and heart disease. Furthermore, obesity has been shown to increase asthma symptoms and frequency of exacerbations.

IL-17 has shown to be upregulated by female sex hormones which may explain the sex specific traits of severe non-Type 2 asthma. In obese mice, IL-17 has shown to be directly responsible for the induction of airway hyperresponsiveness (AHR), thus making it a potential target for treatment. It is especially of interest that none of the previously performed human studies have investigated the effect of blocking IL-17 on AHR. A previous study investigating the effect of blocking IL-17 on lung function, measured as change in FEV1 (forced expiratory volume in 1 second) in moderate to severe patients with asthma, did not find any significant effect. However, this study included both men and women as well as lean and obese participants which could explain the lack of clinical difference. Another previous study also showed no effect of anti-IL17 in general. However, this study showed that those with the greatest reversibility to bronchodilators had the best improvement in symptoms. Although negative, these studies brought us further by showing that anti-IL-17 treatment was safe and tolerable for patients with moderate to severe asthma. Oscillometry has been known for several decades but is only on its' way into clinical practice. Oscillometry is more sensitive than spirometry in detecting small airway disease and AHR. Thus, using oscillometry in studies investigating airway resistance in asthmatic individuals in addition to spirometry, is warranted.

Objectives The overall objective of this study is to determine whether AHR and airway resistance is reduced when initiating treatment with anti-IL17 antibodies for other indications than pulmonary disease. Changes in AHR to methacholine challenge will be reported as response-dose-ratio before and after initiation of anti-IL17. Airway resistance will be assessed using both conventional spirometry for measuring changes in FEV1 and Airwave oscillometry.

Hypothesis

Primary hypothesis: In rheumatologic and dermatological patients commencing anti-IL-17 for other reasons than pulmonary disease, we expect a reduction in airway responsiveness to methacholine challenge after 2-4 months of treatment when compared to prior to initiation of anti-IL-17 treatment.

Secondary hypotheses: Anti-IL17 treatment will show no effect on FEV1, measured using conventional spirometry but will improve measures of airwave oscillometry.

ELIGIBILITY:
Inclusion Criteria:

* Patients planning to start treatment with anti-IL-17 antibodies

Exclusion Criteria:

* Current pregnancy
* FEV1 < 1.5L or less than 60% of predicted value expected.
* Previous anaphylactic shock or severe allergic reaction to medicine
* Uncontrolled hypertension
* Myocardial infarction or stroke within the last 3 months
* Known aortic aneurysm
* Recent eye surgery or risk of elevated intracranial pressure
* Treatment with systemic corticosteroids within 6 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be adult (18 years or older) rheumatologic og dermatologic patients planning to start treatment with anti-IL-17 antibodies. Participants must not have any conditions excluding them from performing a methacholine challenge (Previous anaphylactic shock, current pregnancy, recent cardiac disease, or FEV1 below 1,5L or 60% of expected. Furthermore, patients must not have been treated with systemic corticosteroids within the past 6 weeks.
Sampling Method: Non-Probability Sample
Enrollment: 74 (Estimated)
Dates: Start 2024-08-02 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Airway hyperresponsiveness | approximately 4 months
  Airway responsiveness to methacholine challenge before and after initiation of anti-IL-17 treatment reported as a dose-response-ratio

SECONDARY OUTCOMES:
Airway resistance | approximately 4 months
  Airway resistance will be assessed using both conventional spirometry for measuring changes in FEV1 and Airwave oscillometry

CONTACTS AND LOCATIONS:
Overall Officials: Jonas A Baekdal, MD, Principal Investigator — University hospital, Hvidovre
Locations (1):
- Respiratory Research Unit Hvidovre Department of Respiratory Medicine, Copenhagen University Hospital, Hvidovre, Capital Region, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Mease PJ, McInnes IB, Kirkham B, Kavanaugh A, Rahman P, van der Heijde D, Landewe R, Nash P, Pricop L, Yuan J, Richards HB, Mpofu S; FUTURE 1 Study Group. Secukinumab Inhibition of Interleukin-17A in Patients with Psoriatic Arthritis. N Engl J Med. 2015 Oct;373(14):1329-39. doi: 10.1056/NEJMoa1412679. PMID 26422723
- [Background] Ly K, Smith MP, Thibodeaux Q, Reddy V, Liao W, Bhutani T. Anti IL-17 in psoriasis. Expert Rev Clin Immunol. 2019 Nov;15(11):1185-1194. doi: 10.1080/1744666X.2020.1679625. Epub 2019 Oct 16. PMID 31603358
- [Background] Al Heialy S, Gaudet M, Ramakrishnan RK, Mogas A, Salameh L, Mahboub B, Hamid Q. Contribution of IL-17 in Steroid Hyporesponsiveness in Obese Asthmatics Through Dysregulation of Glucocorticoid Receptors alpha and beta. Front Immunol. 2020 Aug 4;11:1724. doi: 10.3389/fimmu.2020.01724. eCollection 2020. PMID 32849611
- [Background] Agache I, Ciobanu C, Agache C, Anghel M. Increased serum IL-17 is an independent risk factor for severe asthma. Respir Med. 2010 Aug;104(8):1131-7. doi: 10.1016/j.rmed.2010.02.018. Epub 2010 Mar 24. PMID 20338742
- [Background] Peters U, Dixon AE, Forno E. Obesity and asthma. J Allergy Clin Immunol. 2018 Apr;141(4):1169-1179. doi: 10.1016/j.jaci.2018.02.004. PMID 29627041
- [Background] Newcomb DC, Cephus JY, Boswell MG, Fahrenholz JM, Langley EW, Feldman AS, Zhou W, Dulek DE, Goleniewska K, Woodward KB, Sevin CM, Hamilton RG, Kolls JK, Peebles RS Jr. Estrogen and progesterone decrease let-7f microRNA expression and increase IL-23/IL-23 receptor signaling and IL-17A production in patients with severe asthma. J Allergy Clin Immunol. 2015 Oct;136(4):1025-34.e11. doi: 10.1016/j.jaci.2015.05.046. Epub 2015 Aug 1. PMID 26242299
- [Background] Kim HY, Lee HJ, Chang YJ, Pichavant M, Shore SA, Fitzgerald KA, Iwakura Y, Israel E, Bolger K, Faul J, DeKruyff RH, Umetsu DT. Interleukin-17-producing innate lymphoid cells and the NLRP3 inflammasome facilitate obesity-associated airway hyperreactivity. Nat Med. 2014 Jan;20(1):54-61. doi: 10.1038/nm.3423. Epub 2013 Dec 15. PMID 24336249
- [Background] Busse WW, Holgate S, Kerwin E, Chon Y, Feng J, Lin J, Lin SL. Randomized, double-blind, placebo-controlled study of brodalumab, a human anti-IL-17 receptor monoclonal antibody, in moderate to severe asthma. Am J Respir Crit Care Med. 2013 Dec 1;188(11):1294-302. doi: 10.1164/rccm.201212-2318OC. PMID 24200404
- [Background] L. K. A. Lundblad, S. Siddiqui, Y. Bossé, and R. J. Dandurand, "Applications of oscillometry in clinical research and practice," Can. J. Respir. Crit. Care, Sleep Med., vol. 5, no. 1, pp. 54-68, Jan. 2021, doi: 10.1080/24745332.2019.1649607.
- [Background] Abdo M, Kirsten AM, von Mutius E, Kopp M, Hansen G, Rabe KF, Watz H, Trinkmann F, Bahmer T; ALLIANCE study group. Minimal clinically important difference for impulse oscillometry in adults with asthma. Eur Respir J. 2023 May 5;61(5):2201793. doi: 10.1183/13993003.01793-2022. Print 2023 May. PMID 36758985
- [Background] Nicholson PJ. The updated ATS/ERS spirometry technical standards. Occup Med (Lond). 2020 May 27;70(3):146-148. doi: 10.1093/occmed/kqaa030. No abstract available. PMID 32073625
- [Background] Coates AL, Wanger J, Cockcroft DW, Culver BH; Bronchoprovocation Testing Task Force: Kai-Hakon Carlsen; Diamant Z, Gauvreau G, Hall GL, Hallstrand TS, Horvath I, de Jongh FHC, Joos G, Kaminsky DA, Laube BL, Leuppi JD, Sterk PJ. ERS technical standard on bronchial challenge testing: general considerations and performance of methacholine challenge tests. Eur Respir J. 2017 May 1;49(5):1601526. doi: 10.1183/13993003.01526-2016. Print 2017 May. PMID 28461290
- [Background] Parnes JR, Molfino NA, Colice G, Martin U, Corren J, Menzies-Gow A. Targeting TSLP in Asthma. J Asthma Allergy. 2022 Jun 3;15:749-765. doi: 10.2147/JAA.S275039. eCollection 2022. PMID 35685846